CLINICAL TRIAL: NCT00001090
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blinded, Phase I Trial to Evaluate the Safety and Immunogenicity of Live Recombinant Canarypox ALVAC-HIV vCP205, Combined With Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) in Healthy, HIV-1 Uninfected Volunteers
Brief Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blinded, Phase I Trial to Evaluate the Safety and Immunogenicity of Live Recombinant Canarypox ALVAC-HIV vCP205 Combined With GM-CSF in Healthy, HIV-1 Uninfected Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 033; 10582 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Reference Values; Granulocyte-Macrophage Colony-Stimulating Factor; AIDS Vaccines; HIV Seronegativity; Dose-Response Relationship, Immunologic; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections | interventions — sargramostim

INTERVENTIONS:
Biological: APL 400-047
Biological: ALVAC-HIV MN120TMG (vCP205)
Drug: Sargramostim

SUMMARY:
To evaluate the safety and immunogenicity of live recombinant canarypox ALVAC-HIV vCP205 in combination with recombinant human granulocyte-macrophage colony-stimulating factor (GM-CSF) at 80 microg and 250 microg. [AS PER AMENDMENT 4/30/99: To study the safety of following 4 ALVAC immunizations with a nucleic acid gag/pol HIV-1 immunogen (APL-400-047, Wyeth-Lederle). To assess the ability of this sequence of immunization to boost the LTL, T-helper cell, and antibody response.] ALVAC-HIV candidate vaccines have induced HIV-specific CTL responses in more than half of recipients in some protocols. Depending on the HIV-1 gene products expressed by the particular ALVAC-HIV candidate vaccine, volunteers have generated anti-Envelope (vCP125, vCP205, and vCP300), anti-Gag (vCP205 and vCP300), and anti-Nef (vCP300) CTL activity. Although 3 to 4 immunizations with the different ALVAC-HIV experimental vaccines induce anti-HIV-1 neutralizing antibodies in a portion, often the majority, of volunteers, the geometric mean titers of these antibodies are modest, usually less than 50. This study will determine whether there is an increase in the anti-HIV antibody titers when GM-CSF is used as an adjuvant with ALVAC-HIV vCP205 and will also examine the kinetics and magnitude of the HIV-specific CTL response.

DETAILED DESCRIPTION:
ALVAC-HIV candidate vaccines have induced HIV-specific CTL responses in more than half of recipients in some protocols. Depending on the HIV-1 gene products expressed by the particular ALVAC-HIV candidate vaccine, volunteers have generated anti-Envelope (vCP125, vCP205, and vCP300), anti-Gag (vCP205 and vCP300), and anti-Nef (vCP300) CTL activity. Although 3 to 4 immunizations with the different ALVAC-HIV experimental vaccines induce anti-HIV-1 neutralizing antibodies in a portion, often the majority, of volunteers, the geometric mean titers of these antibodies are modest, usually less than 50. This study will determine whether there is an increase in the anti-HIV antibody titers when GM-CSF is used as an adjuvant with ALVAC-HIV vCP205 and will also examine the kinetics and magnitude of the HIV-specific CTL response.

In this randomized, placebo-controlled, double-blinded study volunteers receive ALVAC-HIV vCP205 at 10^6.3 TCID50 or placebo and GM-CSF or placebo by intramuscular injection at Months 0, 1, 3, and 6 as follows:

Group A: vCP205 plus GM-CSF placebo (10 volunteers) Group B: vCP205 plus 80 microg GM-CSF (10 volunteers) Group C: vCP205 plus 250 microg GM-CSF (10 volunteers) Group D: vcP205 placebo plus GM-CSF placebo (6 volunteers). [AS PER AMENDMENT 04/30/99: Boosting with APL-400-047 HIV-1 gag/pol DNA is added for volunteers who have received all scheduled immunization in the original protocol. Volunteers in Groups A, B, and C will receive booster intramuscular injections of DNA vaccine at Months 0 and 1, those in Group D will receive DNA control (bupivacaine carrier alone) at Months 0 and 1].

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Negative ELISA for HIV within 8 weeks prior to immunization.
* CD4 count of 400 cells/mm3 or higher.
* Normal history and physical examination.
* Viable EBV line prior to initial immunization. [AS PER AMENDMENT 4/30/99:
* Negative anti-dsDNA antibodies (for volunteers receiving booster vaccine).]

Exclusion Criteria

Co-existing Condition:

Volunteers with the following conditions or symptoms are excluded:

* Medical or psychiatric condition or occupational responsibilities that preclude compliance with the protocol.
* Recent suicidal ideation or psychosis.
* Active syphilis. NOTE:
* If the serology is documented to be a false positive or due to a remote (greater than 6 months) treated infection, the volunteer is eligible.
* Active tuberculosis. NOTE:
* Volunteers who have a positive PPD and a normal chest x-ray showing no evidence of TB and who do not require INH therapy are eligible.
* Positive for hepatitis C antibody or hepatitis B surface antigen.
* Allergy to eggs, neomycin, or thimerosal. [AS PER AMENDMENT 4/30/99:
* Hypersensitivity to bupivacaine or other amide-type anesthetics (e.g., lidocaine, mepivacaine) for volunteers receiving booster vaccine).]

Concurrent Medication:

Excluded:

Lithium or cimetidine.

Volunteers with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, or autoimmune disease.
* History of cancer unless there has been surgical excision with reasonable assurance of cure.
* History of suicide attempts or past psychosis.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance requiring hospitalization or emergent care (e.g., Stevens-Johnson syndrome, bronchospasm, or hypotension).

[AS PER AMENDMENT 11/13/97:

* History of cardiac disease or cardiac arrhythmias.]

Prior Medication:

Excluded:

* Live attenuated vaccines within 60 days of study. NOTE:
* Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary, but should be given at least 2 weeks away from HIV immunizations.
* Experimental agents within 30 days prior to study.
* Blood products or immunoglobulin in the past 6 months.
* HIV-1 vaccines or placebo as part of a previous HIV vaccine trial.
* Immunosuppressive medications.

Risk Behavior:

Excluded:

Volunteers with an identifiable higher-risk behavior for HIV infection (i.e., AVEG Risk Group C or D), including a history of injection drug use within 12 months prior to enrollment or higher-risk sexual behavior as defined by the AVEG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Study Completion 1999-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: T Evans, Study Chair
Locations (4):
- United States (4):
  - UAB AVEG, Birmingham, Alabama
  - JHU AVEG, Baltimore, Maryland
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee